CLINICAL TRIAL: NCT04635891
Title: Motor Outcomes to Validate Evaluations in FSHD (MOVE FSHD)
Acronym: MOVE FSHD
Status: Recruiting | Type: Observational
Sponsor: University of Kansas Medical Center (Other)
Collaborators: FSHD Society, Inc. (Unknown); Friends Research Institute, Inc. (Other); University of Rochester (Other); University of Nevada, Reno (Other); FSHD Canada (Unknown); Avidity Biosciences, Inc. (Industry); AMRA Medical (Unknown); Seattle Children's Hospital (Other); Dyne Therapeutics (Industry); Hoffmann-La Roche (Industry); Springbok Analytics (Unknown)
Responsible Party: Sponsor
Other Study IDs: STUDY00145405
Record Dates: First submitted 2020-10-29; First posted 2020-11-19 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: FSHD

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Saliva samples that are collected will be sent to University of Nevada Reno for DNA methylation testing, and participants will receive results. DNA, RNA, plasma, and serum biomarker samples that are collected will be sent to University of Rochester Medical Center and will be stored in a biorepository for future research. Muscle tissue samples that are collected will be sent for RNA sequencing and commercial assay validation. Remaining muscle tissue will be sent to University of Rochester Medical Center biorepository for future research use.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- MOVE FSHD Study Visits: Patients will receive standard of care as determined by their treating physician. Study visits will occur per standard of care and are anticipated to occur at least once a year.

SUMMARY:
The primary goal of this proposal is to collect motor and functional outcomes specific to FSHD over time. By collecting measures specific to FSHD, this will help ensure the best level of clinical care is being provided. Also, the hope is to speed up drug development by gaining a better understanding of how having FSHD impacts motor function and other health outcomes (i.e. breathing, wheelchair use, etc.) and how big a change in motor function would be clinically meaningful to those with FSHD.

Motor Outcomes to Validate Evaluations in FSHD (MOVE FSHD) will have approximately 450 FSHD participants followed for a minimum of 3 years. A subset of MOVE FSHD participants, approximately 200, will participate in the MOVE+ sub-study which includes whole body MRI and reachable workspace, as well as optional muscle biopsy and wearable device (US participants only).

ELIGIBILITY:
Inclusion Criteria:

* Genetically confirmed FSHD (types 1 or 2) or clinical diagnosis of FSHD with characteristic findings on exam and an affected parent or offspring.

Exclusion Criteria:

* Unwilling or unable to provide informed consent.
* Any other medical condition which in the opinion of the investigator would interfere with study participation.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants with FSHD that are seen in the researchers clinic.
  This study is meant to be 'inclusive' and cover the full range of clinical FSHD: including children and adults, all ranges of abilities (ambulatory and non-ambulatory), and both genetic types of FSHD.
Sampling Method: Non-Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2020-12-15 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
10m walk/run | Baseline - 5 years
  The 10-meter walk/run (previously the 30 foot go) or gait speed task will be performed during study visits. This task tests a range of different abilities, from power, to endurance, and balance. Also, the 10 meter walk/run is a predictor of loss of ambulation in Duchenne Muscular Dystrophy.
Shoulder and Arm Range of Motion | Baseline - 5 years
  Range of motion tasks mimicking lifting or reaching up will be performed.
Shoulder and Arm Function | Baseline - 5 years
  Participants will be timed on stacking cans.
Spirometry (FVC, FEV1, PCF) | Baseline - 5 years
  Investigators will obtain forced vital capacity and forced expiratory volume in 1 second, both standardized outcomes used commonly in clinic and clinical trials. Also, for sites who routinely collect Peak Cough Flow this will also be obtained.

SECONDARY OUTCOMES:
Trunk Function | Baseline - 5 years
  There are no specific functional tasks designed to measure trunk function in FSHD so Investigators have chosen a practical task that will reflect changes in core truncal muscle groups. The ability to sit up and the timed supine to sitting test reflects core muscle strength and coordination.
Hand Function | Baseline - 5 years
  Hand function is captured by examining hand grip strength.
Timed Up and Go (TUG) | Baseline - 5 years
  Balance and mobility are assessed by using the Timed Up and Go (TUG), a standard outcome measure for the elderly that is also increasingly being used in neuromuscular disorders. Participants are asked to rise from a chair, walk 3 meters, turn 180 degrees and return to a seated position in the chair.
Saliva Methylation | Baseline (collected only once)
  Investigators will isolate DNA from blood cells in saliva - and will determine the methylation levels in the 4q region on chromosome 4 using this new technique. Investigators will compare methylation levels between participants and compare to other clinical information collected in this study.
FSHD Clinical Severity Scores | Baseline - 5 years
  A limited physical exam and strength testing will be used to derive two FSHD clinical severity scores. These severity scores both rank weakness in the face, shoulders, arms, distal, and proximal lower extremities on either a 10 or 15 point scale. The higher the severity score the more affected the individual.
Patient-Reported Outcomes Measurement Information System-57 (PROMIS57) | Baseline - 5 years
  The PROMIS57 is an instrument developed by the NIH which generates scores for physical function, and the impact of physical limitations on daily life. 57 questions are summed into a total score, which is transformed into a normalized t-score with 50 representing normal, and lower scores representing increasing disability.
The Upper Extremity Functional Index | Baseline - 5 years
  This index measures upper extremity dysfunction. 20 questions are combined into a total score, the score is transformed into a normalized score with 80 representing normal, and lower scores representing increasing disability.
Exercise and Pain Assessment | Baseline - 5 years
  An exercise and pain assessment questionnaire was comprised specifically for this study and will be completed at every visit.
The Facial Disability Index (FDI) | Baseline - 5 years
  The FDI is a short 5 item questionnaire. The five questions are summed into total score which transformed onto a percentage scale, with 100 representing normal, and lower scores representing increasing disability.
FSHD Rasch-built overall disability scales (FSHD-RODS) | Baseline - 5 years
  The FSHD-RODS is a questionnaire about the relationship between daily activities and health. 32 questions are are constructed using a modern clinimetric technique, the Rasch analysis, which by ordering the items in increasing difficulty, allows for the calculation of the sum of item scores to achieve a total score. Answers provide information about how FSHD affects daily and social activities and to what degree participants are able to perform usual activities.
MIP/MEP and SNIP | Baseline - 5 years
  For sites who routinely obtain negative inspiratory or expiratory force (MIP/MEP) will be collected.
4 Stair Climb | Baseline - 5 years
  Time to ascend and descend 4 standard stairs.
Manual Muscle Testing (MMT) | Baseline - 5 years
  For MMT a modified Medical Research Council 13-point scale will be used - with standardized positions for each muscle.

OTHER OUTCOMES:
Biospecimen Retention: Samples with DNA, RNA, plasma, and serum | Baseline - 5 years
  Optional sub-study collecting DNA, RNA, plasma, and serum for biobanking.
Remote Assessment Pilot | Baseline - 5 years
  A sub-group of approximately 20 participants will perform remote assessments in the home. The remote assessments are meant to capture the assessments that occur during a routine in-person visit, and will overlap functional categories, to include reaching and lifting objects, core functional measures, measures of gait and balance, and midarm and hand tasks. Measures of respiratory (FVC, FEV1, PCF, SNIP), bulbar function, and handgrip strength will also be included. Functional measures will be modified to allow for independent and/or via two-way video performance.
MRI | Baseline - 12-Month
  Whole body MRI will be performed for a sub-group of approximately 200 participants. MRI is recognized as a gold standard for body composition analysis, enabling a more complete description of a person's body composition profile from a single examination.In addition, we will include analysis to help make needle biopsy based on STIR and quantitative fat fraction more efficient with higher yield using standard fiducial markings and body landmarks.
Muscle Biopsy | Baseline - 4-Month
  Muscle biopsy will be performed for a sub-group of approximately 200 participants. Muscle biopsies will be performed at the baseline visit and for a subset of 20 participants at 4 months. We will use MRI analysis to help inform which lower extremity muscle will be chosen for biopsy. Muscle samples will be used to recapitulate RNA sequencing to confirm prior DUX4 target selection. In addition, other early or late genes of interest may be included which are FSHD-related but not specific to DUX4. We will also select 4 control genes for quality assurance, 2 to confirm muscle tissue, and 2 to rule out high fat content.
Reachable and Functional Workspace | Baseline - 24-Months
  Reachable and Functional Workspace will be performed for a sub-group of approximately 200 participants. Participants are seated in front of a stereo-camera and perform a standardized upper extremity movement protocol under the supervision of a study clinical evaluator. Five-hundred-gram wrist weights will be added. The standardized simple set of movements consist of lifting the arm from the resting position to above the head while keeping the elbow extended, performing the same movement in vertical planes at around 0, 45, 90, 135 degrees. The second set of movements consists of horizontal sweeps at the level of the umbilicus and shoulder. Each set of movements is repeated three times for left and right arm.
Syde Wearable Device | Baseline - 24-Months
  The purpose of the wearable device is to accurately measure upper and lower limb movement during normal daily living. In FSHD, muscles are affected asymmetrically, therefore, measurements with the wearable device will be taken from the upper and lower limbs bilaterally.
Motor Function Measure 32 (MFM32) | Baseline - 24-months (remote assessment and MOVE+ peds pilot only)
  32-item Motor Function Measure (MFM32) is a clinician-reported outcome measure used to assess the functional abilities of individuals with neuromuscular diseases.
FSHD COM Peds | Baseline - 24-Months
  We will collect the FSH-Composite outcome measure for children and adolescents. As with the FSHD-COM, the body regions assessed match areas of importance identified by patients and include leg function; shoulder and arm function; trunk function, hand function; and functional balance. The FSHD-COM Peds was modified by adding lighter weights to the shoulder abduction and flexion and elbow flexion items to accommodate motor development and lower strength levels seen in children. Most of the items are scored on a 5-point ordinal scale (0 = normal/not affected and 4= being severely affected or unable to complete the item) with the exception of the shoulder abduction/flexion and elbow flexion items which have been expanded and are scored on a 7-point scale using the additional weight categories. Thus, the total score for the FSHD-COM Peds is 84 (compared to 72 for the FSHD-COM).

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Statland, MD, Principal Investigator — University of Kansas Medical Center; Rabi Tawil, MD, Principal Investigator — University of Rochester
Locations (20):
- United States (15):
  - David Geffen School of Medicine at UCLA, Los Angeles, California
  - Neuromuscular Disorders Program at Stanford University School of Medicine, Stanford, California
  - University of Colorado Anschutz Medical Campus, Aurora, Colorado
  - Univeristy of Florida Gainesville, Gainesville, Florida
  - University of Iowa, Iowa City, Iowa
  - Univeristy of Kansas Medical Center, Kansas City, Kansas
  - Kennedy Krieger Institute, Baltimore, Maryland
  - University of Rochester Medical Center, Rochester, New York
  - The Ohio State University Medical Center, Columbus, Ohio
  - Austin Neuromuscular Center, Austin, Texas
  - Univeristy of Texas Southwestern Medical Center, Dallas, Texas
  - University of Texas Health San Antonio, San Antonio, Texas
  - University of Utah, Salt Lake City, Utah
  - Virginia Commonwealth University, Richmond, Virginia
  - University of Washington Medical Center, Seattle, Washington
- University of Sao Paulo, São Paulo, Brazil
- Canada (3):
  - University of Calgary, Calgary, Alberta
  - Ottawa Hospital Research Institute, Ottawa, Ontario
  - University of McGill, Montreal, Quebec
- Sheffield Teaching Hospital, Sheffield, South Yorkshire, United Kingdom